CLINICAL TRIAL: NCT02467933
Title: The Effect of Informative Letters on the Prescription and Receipt of Seroquel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); General Services Administration (GSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JPAL-LETTERS-SEROQUEL
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Economics; Fraud; Delivery of Health Care; Health Expenditures; Centers for Medicare and Medicaid Services (U.S.)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo arm receives a placebo letter unrelated to Seroquel
  Interventions: Other: Placebo letter
- Informative Letter (Experimental): The interventional arm prescribers receive an initial informative letter (called a comparative billing report or peer activity report) followed by 2 followup informative letters at approximately 3 month intervals.
  Interventions: Other: Initial Informative letter; Other: Followup Informative Letter

INTERVENTIONS:
Other: Placebo letter — The placebo letter describes a new rule in Medicare that requires prescribers to enroll in Medicare
  Arms: Placebo
Other: Initial Informative letter — The intervention is a letter that describes the Seroquel prescribing activity of the individual in comparison to a peer group of similar prescribers. It highlights the fact that the prescriber's activity is highly unlike her peers.
  Arms: Informative Letter
Other: Followup Informative Letter — The followup informative letter is identical to the initial informative letter except it provides an update on more recent prescribing rather than a description of earlier prescribing.
  Arms: Informative Letter

SUMMARY:
Abusive prescribing exposes patients to unnecessary health risks and results in wasteful public expenditures. This study will evaluate an innovative approach to fighting abusive prescription: sending letters to suspected inappropriate prescribers warning them that they are outliers compared to their peers and have been flagged for review. The study will target high prescribers of Seroquel (Quetiapine), an atypical antipsychotic. Using claims data, the investigators will assess the effect of the letters on prescribing of Seroquel, receipt of Seroquel by patients, substitution behavior by prescribers and patients, and health outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* General care practitioner
* Outlier with respect to the count of Seroquel prescription drug treatments relative to peer group of prescribers in 2013 and 2014
* Outlier with respect to the count of Seroquel 30-day equivalent prescription drug treatments relative to peer group of prescribers in 2013 and 2014

Exclusion Criteria:

* Deceased

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5055 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
30-day equivalent prescribing of Seroquel treatments | 9 months
  The prescribing of Seroquel over the 9 months following the initial sending of the letters. Prescribing is defined as the total "days supply" of Seroquel attributed to the prescriber, expressed in "30-day equivalents" i.e. divided by 30.

SECONDARY OUTCOMES:
30-day equivalent prescribing of Seroquel treatments | 3 months
30-day equivalent prescribing of Seroquel treatments | 6 months
30-day equivalent prescribing of Seroquel treatments | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sacarny, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sacarny A, Barnett ML, Le J, Tetkoski F, Yokum D, Agrawal S. Effect of Peer Comparison Letters for High-Volume Primary Care Prescribers of Quetiapine in Older and Disabled Adults: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Oct 1;75(10):1003-1011. doi: 10.1001/jamapsychiatry.2018.1867. PMID 30073273
- See also: American Economic Association Randomized Controlled Trials Registry Entry — https://www.socialscienceregistry.org/trials/729
- Available data/document: Study Protocol: 449 — https://www.socialscienceregistry.org/trials/729 — Study protocol archived on American Economic Association Social Science Registry page.
- Available data/document: Statistical Analysis Plan: 448 — https://www.socialscienceregistry.org/trials/729 — Pre-specified analysis plan archived on American Economic Association Social Science Registry page. Final version prior to unblinding: Version 2.0 (March 5, 2016)